CLINICAL TRIAL: NCT06289777
Title: Aortic Remodeling After Endovascular Management of Type B Aortic Dissection.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed hesham abdelrahem husiein, Assistant lecturer, Assiut University
Other Study IDs: aortic remodeling
Record Dates: First submitted 2024-02-17; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Type B Aortic Dissection
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TEVAR — minimally invasive endovascular intervention to treat aortic dissection

SUMMARY:
Assess the clinical outcome, morphological changes and behaviour of type B aortic dissection after endovascular repair.

DETAILED DESCRIPTION:
Aortic dissection (AD) is considered the most common catastrophic event of the aorta, and its incidence has been reported to be ≈3/100000 per year, exceeding that of ruptured abdominal aortic aneurysm.

AD is a dynamic process and can occur anywhere along the course of the aorta, with the pathognomonic lesion being an intimal tear followed by blood surging either antegrade (typically) or retrograde, cleaving the the intima and medial layers of the aortic wall longitudinally for a variable distance, thus creating a true and false lumens.

Aortic dissections are classified by chronicity, anatomic location of false lumen, generally the entry tear and longitudinal extent, and the presence or absence of complicating features.

Temporally, AD is categorized as acute phase {<14 days}, subacute {15-90 days}, and chronic {>90 days}.

Thoracic Endovascular Aortic Repair (TEVAR) has emerged as the first-line therapy for the treatment of AD, with better short-term results than open repair due to a significant decrease in perioperative morbidity and mortality.

By covering the primary entry tear with stent-grafts, the blood flow is redirected into the true lumen, resolving malperfusion and/or preventing rupture of the false lumen, followed by its regression and re-expansion of the true lumen, which is known as "Aortic remodeling"

ELIGIBILITY:
Inclusion Criteria:

1. Complicated Stanford type B dissections:

   * Rupture.
   * malperfusion (visceral, extremities or spinal cord ischemia).
2. High-risk aortic dissections:

   * Refractory pain, refractory hypertension or bloody pleural effusion.
   * High-risk radiographic features (max. aortic diameter >40mm, false lumen diameter >22mm, 1ry entry tear >1cm, entry tear location on the lesser curve and radiographic only malperfusin).
3. Aortic anatomy suitable for stent graft therapy:

   * Proximal landing zone (diameters between 15 and 42mm, measured form outer wall to outer wall) isn't aneurysmal, dissected or significantly thrombosed.
   * Proximal landing zone length ≥20mm.
   * Radius of curvature ≥20mm for aortic arch landing zones.
   * Arch or distal aortic angulation 45≤ degrees.
4. Compatible Iliac and/or femoral access vessel morphology (diameter and tortousity) that allows endovascular access to the dissection site with the delivery system of the appropriately sized device, with or without the use of either surigcal or endovascular conduit.
5. Age ≥18yrs.
6. Life expectancy >2yrs

Exclusion Criteria:

1. Known hypersensitivity to device component or contraindication to anticoagulation or contrast media.
2. Systemic or local infection that may increase the risk of endovascular graft infection.
3. Subjects with past descending or abdominal aortic interventions.
4. Un-correctable coagulopathy
5. Active vasculitis
6. Inability or refusal to give informed consent by subject or legal representative
7. Subject is unwilling to comply with the follow-up schedule.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: complicated or high-risk acute, subacute or chronic type B aortic dissection.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of aortic remodeling | 2 years
  evaluation of diameter changes between the preoperative and postoperative CTs measurements in millimetres . The true lumen index (Tli) is calcuated by dividing thr true lumen diameter by the whole lumen (transaortic) diameter. The fasle lumen index (Fli) is calculated in the same manner. The desirable TLi value approaches or equals 1 (suggesting increase in true lumen to normal), whereas the sought-after FLi value approaches or equals 0 (suggesting shrinkage in false lumen).
technical success | baseline
  successful delivery and deployment of the device with coverage of the 1ry tear at implant with no detected endoleak on angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

REFERENCES:
- [Background] Watanabe Y, Shimamura K, Yoshida T, Daimon T, Shirakawa Y, Torikai K, Sakamoto T, Shijo T, Toda K, Kuratani T, Sawa Y. Aortic remodeling as a prognostic factor for late aortic events after thoracic endovascular aortic repair in type B aortic dissection with patent false lumen. J Endovasc Ther. 2014 Aug;21(4):517-25. doi: 10.1583/13-4646R.1. PMID 25101579
- [Background] Hagedorn MN, Meisenbacher K, Skrypnik D, Bischoff MS, Bockler D. Standing the test of time: total aortic remodeling 13 years after TEVAR for acute type B aortic dissection. Indian J Thorac Cardiovasc Surg. 2024 Jan;40(1):86-90. doi: 10.1007/s12055-023-01586-5. Epub 2023 Sep 4. PMID 38125333
- [Background] Rodriguez JA, Olsen DM, Lucas L, Wheatley G, Ramaiah V, Diethrich EB. Aortic remodeling after endografting of thoracoabdominal aortic dissection. J Vasc Surg. 2008 Jun;47(6):1188-94. doi: 10.1016/j.jvs.2008.01.022. Epub 2008 Apr 28. PMID 18440180
- [Background] Lombardi JV, Cambria RP, Nienaber CA, Chiesa R, Mossop P, Haulon S, Zhou Q, Jia F; STABLE investigators. Aortic remodeling after endovascular treatment of complicated type B aortic dissection with the use of a composite device design. J Vasc Surg. 2014 Jun;59(6):1544-54. doi: 10.1016/j.jvs.2013.12.038. Epub 2014 Feb 19. PMID 24560244
- [Background] Riambau V, Bockler D, Brunkwall J, Cao P, Chiesa R, Coppi G, Czerny M, Fraedrich G, Haulon S, Jacobs MJ, Lachat ML, Moll FL, Setacci C, Taylor PR, Thompson M, Trimarchi S, Verhagen HJ, Verhoeven EL, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus ES, Hinchliffe RJ, Kakkos S, Koncar I, Lindholt JS, Vega de Ceniga M, Vermassen F, Verzini F, Document Reviewers, Kolh P, Black JH 3rd, Busund R, Bjorck M, Dake M, Dick F, Eggebrecht H, Evangelista A, Grabenwoger M, Milner R, Naylor AR, Ricco JB, Rousseau H, Schmidli J. Editor's Choice - Management of Descending Thoracic Aorta Diseases: Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2017 Jan;53(1):4-52. doi: 10.1016/j.ejvs.2016.06.005. No abstract available. PMID 28081802
- [Background] Iannuzzi JC, Stapleton SM, Bababekov YJ, Chang D, Lancaster RT, Conrad MF, Cambria RP, Patel VI. Favorable impact of thoracic endovascular aortic repair on survival of patients with acute uncomplicated type B aortic dissection. J Vasc Surg. 2018 Dec;68(6):1649-1655. doi: 10.1016/j.jvs.2018.04.034. Epub 2018 Jun 15. PMID 29914833
- [Background] Jiang X, Liu Y, Zou L, Chen B, Jiang J, Fu W, Dong Z. Long-Term Outcomes of Chronic Type B Aortic Dissection Treated by Thoracic Endovascular Aortic Repair. J Am Heart Assoc. 2023 Jan 3;12(1):e026914. doi: 10.1161/JAHA.122.026914. Epub 2022 Nov 16. PMID 36382952
- [Background] Lombardi JV, Hughes GC, Appoo JJ, Bavaria JE, Beck AW, Cambria RP, Charlton-Ouw K, Eslami MH, Kim KM, Leshnower BG, Maldonado T, Reece TB, Wang GJ. Society for Vascular Surgery (SVS) and Society of Thoracic Surgeons (STS) Reporting Standards for Type B Aortic Dissections. Ann Thorac Surg. 2020 Mar;109(3):959-981. doi: 10.1016/j.athoracsur.2019.10.005. Epub 2020 Jan 27. PMID 32000979
- [Background] Sobocinski J, Lombardi JV, Dias NV, Berger L, Zhou Q, Jia F, Resch T, Haulon S. Volume analysis of true and false lumens in acute complicated type B aortic dissections after thoracic endovascular aortic repair with stent grafts alone or with a composite device design. J Vasc Surg. 2016 May;63(5):1216-24. doi: 10.1016/j.jvs.2015.11.037. Epub 2016 Jan 22. PMID 26806523
- [Background] Trimarchi S, Gleason TG, Brinster DR, Bismuth J, Bossone E, Sundt TM, Montgomery DG, Pai CW, Bissacco D, de Beaufort HWL, Bavaria JE, Mussa F, Bekeredjian R, Schermerhorn M, Pacini D, Myrmel T, Ouzounian M, Korach A, Chen EP, Coselli JS, Eagle KA, Patel HJ. Editor's Choice - Trends in Management and Outcomes of Type B Aortic Dissection: A Report From the International Registry of Aortic Dissection. Eur J Vasc Endovasc Surg. 2023 Dec;66(6):775-782. doi: 10.1016/j.ejvs.2023.05.015. Epub 2023 May 16. PMID 37201718